CLINICAL TRIAL: NCT06873464
Title: Evaluation of the Efficacy of Transcranial Direct Current Stimulation in Reducing Fatigue and Improving Quality of Life in Patients With Multiple Sclerosis: A Randomized Clinical Trial
Acronym: tDCS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Marina Castel Sánchez, Marina Castel Sánchez, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIm25-10
Record Dates: First submitted 2025-02-20; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis, MS
Keywords: Transcranial Direct-Current Stimulation; fatigue; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three cycles of tDCS combined with motor tasks group (Experimental): Three 2-week cycles. Each cycle includes tDCS combined with motor tasks. The initial session of the first cycle and the final sessions of the second and third cycles last 45 minutes, involving tDCS and motor tasks, and MFIS, MSQOL-54, and BBS assessments. Other sessions last 30 minutes, focusing on tDCS and motor tasks.
  tDCS Parameters: Intensity: 2000 mA Application Time: 20 minutes with a 10-second ramp-up Electrode placement: Anode at C3, Cathode at FP2
  Interventions: Other: Three cycles of tDCS combined with motor tasks
- Two cycles of tDCS combined with motor tasks group (Active Comparator): Two 2-week tDCS cycles will be conducted. Each cycle includes tDCS combined with motor tasks. The initial session of the first cycle and the final sessions of the second cycle last 45 minutes, involving tDCS and motor tasks, and MFIS, MSQOL-54, and BBS assessments. Other sessions last 30 minutes, focusing on tDCS and motor tasks.
  tDCS Parameters:
  * Intensity: 2000 mA
  * Time: 20 minutes with a 10-second ramp-up
  * Electrode Placement: Anode at C3, Cathode at FP2
  Interventions: Other: Two cycles of tDCS combined with motor tasks

INTERVENTIONS:
Other: Three cycles of tDCS combined with motor tasks — Three cycles of 2 weeks duration each combining tDCS and motor task.
  Initial Assessment (V0): Collect demographic data and EDSS, MFIS, MSQOL-54, and BBS results.
  First Cycle: 2 weeks, Monday to Friday, with a weekend break. Post-First Cycle Assessment (V1): Reassess MFIS, MSQOL-54, and BBS. Washout Period: 1 month without tDCS. Second Cycle: 2 weeks, Monday to Friday, with a weekend break. Final Assessment after Second Cycle (V2): Reassess MFIS, MSQOL-54, and BBS. Washout Period: 1 month. Third Cycle: 2 weeks. Final Assessment after Third Cycle (V3): Reassess MFIS, MSQOL-54, and BBS.
  Arms: Three cycles of tDCS combined with motor tasks group
Other: Two cycles of tDCS combined with motor tasks — Initial assessment (V0): Prior to the first tDCS cycle, demographic data and results from the EDSS, MFIS, MSQOL-54, and BBS scales will be collected.
  First cycle: 2 weeks Post-first cycle assessment (V1): Reassess MFIS, MSQOL-54, and BBS scales. Washout period: 1 month without tDCS treatment. Second cycle: 2 weeks, with sessions from Monday to Friday and a weekend break. Final assessment (V2): After the second cycle, reassess MFIS, MSQOL-54, and BBS scales.
  Follow-up assessment (V3): 45 days after treatment completion.
  Arms: Two cycles of tDCS combined with motor tasks group

SUMMARY:
The goal of this clinical trial is to evaluate whether the application of three 2-week cycles of tDCS combined with motor therapy is more effective in reducing fatigue in adult patients with multiple sclerosis, compared to the application of two cycles of the same treatment. The main questions aim to answer:

* Is the application of three 2-week cycles of tDCS combined with motor therapy (experimental group) more effective for the recovery of fatigue in adult patients with multiple sclerosis compared to the application of two cycles of the same treatment (control group)?
* Is tDCS combined with motor therapy effective in improving fatigue in adult patients with multiple sclerosis in both study arms, i.e., in the pre-post assessment of the experimental group and the pre-post assessment of the control group? Researchers will compare the application of three 2-week cycles of tDCS combined with motor therapy (experimental group) to the application of two cycles of the same treatment (control group) to see if the experimental group shows greater recovery of fatigue in adult patients with multiple sclerosis.

Participants will:

* Visit the clinic for two weeks to be evaluated (baseline measurement and first post-treatment assessment) and receive the first cycle of treatment from Monday to Friday.
* Have a washout period of one month between the first and the second cycle.
* Visit the clinic for two weeks to receive the second cycle of treatment and be evaluated (second post-treatment assessment).
* Only participants in the experimental group will have another washout period of one month and visit the clinic to receive a third cycle of treatment and to be evaluated (third post-treatment assessment).
* Only participants in the control group will visit the clinic one and a half months after completing their second cycle to be measured as a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis defined according to the McDonald criteria (2017 revised version).
* Age between 18 and 75 years.
* No relapse in the last 2 months.
* Fatigue experienced in the last 6 months, according to the Fatigue Severity Scale (FSS > 4).

Exclusion Criteria:

* Patients who have not had stable pharmacological treatment in the last month.
* Patients with contraindications to the use of tDCS, such as: defibrillator, pacemaker, brain stimulator, implanted intracranial metals, skull fractures or fissures, damaged skin or recent scars, epilepsy, pregnancy.
* Patients who are undergoing or need to undergo immunosuppressive treatment for MS with Ocrelizumab, Rituximab, Lemtrada, or Mavenclad one week before or during the application of tDCS.
* Patients with cognitive difficulties that prevent them from understanding the applied scales.
* Patients who experience adverse effects from tDCS treatment.
* Inability to remain in the study and complete the third cycle and/or the V3 assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue Impact | Assessed at baseline (V0), after 2 weeks (V1), after 6 weeks (V2), and after 14 weeks (V3).
  Fatigue Impact Scale measures the impact of fatigue on daily functioning across three domains: cognitive, physical, and psychosocial. It consists of 40 items rated on a scale from 0 (no problem) to 4 (extreme problem). The total score ranges from 0 to 160, with higher scores indicating greater fatigue impact. Subscale scores are also calculated for each domain

SECONDARY OUTCOMES:
Multiple Sclerosis Quality of Life assessment | Assessed at baseline (V0), after 2 weeks (V1), after 6 weeks (V2), and after 14 weeks (V3)
  Multiple Sclerosis Quality of Life - 54 (MSQOL-54) is a multidimensional health-related quality of life measure combining generic and MS-specific items. It includes 54 items generating 12 subscales and two summary scores (physical and mental health). There is no single overall score. Subscale scores and summary scores are derived from a weighted combination of scale scores. Higher scores indicate better quality of life
Balance | Assessed at baseline (V0), post-first cycle (V1, after 2 weeks), post-second cycle (V2, after 6 weeks), and post-third cycle (V3, after 14 weeks)).
  The Berg Balance Scale assesses static balance and fall risk through 14 tasks, each scored from 0 (lowest function) to 4 (highest function). The total score ranges from 0 to 56. Scores below 45 indicate a higher risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Esclerosis Multiple Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided